CLINICAL TRIAL: NCT05469867
Title: A Single Arm, Pivotal, Open Label, Multi-centre Clinical Investigation to Evaluate the Clinical Safety and Performance of the CorNeat EverPatch, A Synthetic Tissue Substitute for Concealment of Artificial Ocular Implants
Brief Title: Pivotal Trial for a Synthetic Tissue Substitute for Concealment of Artificial Ocular Implants
Acronym: EverPatch
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to stop the trial due to a shift in strategic business priorities.
Sponsor: CorNeat Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DMS-34948
Record Dates: First submitted 2022-07-18; First posted 2022-07-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Glaucoma Eye; Tissue Breakdown

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corneat EverPatch - Synthetic Tissue Substitute for Covering Ophthalmic Implants (Experimental)
  Interventions: Device: CorNeat EverPatch

INTERVENTIONS:
Device: CorNeat EverPatch — The CorNeat EverPatch will be implanted subconjunctivally over an ocular implant (e.g. glaucoma shunt, exposed suture tags) and fixed to the eye wall. The overlying conjunctiva will be closed over the patch.

SUMMARY:
This clinical trial will assess the clinical safety and performance of the CorNeat EverPatch device used as a tissue substitute for concealment of artificial ocular implants.

DETAILED DESCRIPTION:
A single arm, pivotal, open label, multi-centre clinical investigation to evaluate the clinical safety and performance of the CorNeat EverPatch, a synthetic tissue substitute for concealment of artificial ocular implants.

Subjects will sign a consent form and will be assessed for eligibility based on clinical examinations and medical history. Upon eligibility verification, subjects will be implanted with the investigational device as part of an ophthalmic surgery in which a concealment of an artificial implant is required. Clinical examinations at follow up will include slit lamp biomicroscopy, assessment of visual acuity and intra ocular pressure, and recording of concomitant medications and any safety issues. Follow up visits will be performed at 1 week, 1-, 2-, 3-, 6-, 9- and 12-months post-op.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged ≥ 18 and ≤ 80 years on screening day
3. Concealment of glaucoma tube shunt or suture tags is indicated
4. Patients with viable and intact conjunctiva
5. Candidates must have the ability and willingness to provide a written informed consent, attend all scheduled visits and comply with study procedures
6. Adequate tear film and lid function as indicated by Tear Film Breakup Time test - more than 5 seconds
7. Visual acuity of light perception or better
8. Female patients of childbearing age must agree to use an acceptable and effective method of contraception throughout the study, including the follow-up period, and have negative pregnancy test at screening.

Exclusion Criteria:

1. Current retinal detachment
2. Active ocular or orbital infection
3. History or evidence of severe inflammatory eye diseases (i.e. uveitis, retinitis, scleritis) in one or both eyes within 6 months prior to planned implantation
4. History of ocular or periocular malignancy
5. History of extensive keloid formation
6. Any known intolerance or hypersensitivity to topical anesthetics, mydriatics, or component of the device, specifically Oxybuprocaine hydrochloride, lidocaine, tropicamide, epinephrine, Iodine solution & aromatic polycarbonate urethane
7. Signs of current infection, including fever and current treatment with antibiotics
8. Severe generalized disease that results in a life expectancy shorter than a year
9. Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
10. Pregnant or breastfeeding female subjects
11. Participation in any study involving an investigational drug or device within 30 days of the study or 5 half-lives of the drug (whichever longer) or ongoing participation in a study with an investigational drug or device
12. Any traumatic perforation of the globe OR tissue gaps/weaknesses, resulting either from traumatic, disease- related or iatrogenic damage OR loss of scleral integrity where use of tissue or substitutes is indicated
13. Vulnerable populations
14. Active drug or alcohol abuse or dependence that, in the opinion of the principle investigator, would interfere with adherence to study requirements
15. Subjects with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (e.g. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive heart failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, uncompensated cirrhosis, active upper GI tract ulceration, active inflammatory disease, malignancy under active treatment)
16. Subjects who receive anti-coagulation treatment which cannot be interfered during the perioperative period
17. Hemoglobin A1C (HbA1c) higher than 8% at screening indicating unbalanced diabetes and/or target organ damage associated with diabetes
18. Subjects receiving chronic systemic immunosuppressants (e.g. steroids, cyclosporine etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | Up to 12 months
  The frequency of all Unanticipated Adverse Device-related Events (UADE) during and following implantation will be recorded

SECONDARY OUTCOMES:
Performance Assessment | 6 & 12 months post-op.
  Tube or suture exposure will be detected by slit-lamp Biomicroscopy throughout the entire follow up period and incidence will be calculated. Prevention of tube or suture exposure associated with conjunctival erosion and graft melting should be demonstrated in at least 90% of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- DaVinci Eye Care, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No